CLINICAL TRIAL: NCT02022020
Title: An Observational Study Assessing the Management of Gastrointestinal and Urogenital Bleeding Events in Patients With Atrial Fibrillation Treated With Dabigatran Etexilate
Brief Title: Management of Gastrointestinal and Urogenital (GI/GU) Bleedings in Atrial Fibrillation Patients Using Pradaxa
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.162
Record Dates: First submitted 2013-11-25; First posted 2013-12-27 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
This study is being conducted to collect data on the management of gastrointestinal and urogenital bleeding events occurring in patients with atrial fibrillation taking dabigatran etexilate.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* >=18 years of age;
* Confirmed diagnosis of Atrial Fibrillation (AF);
* Documentation that the patient had an acute GI and/or GU bleeding event and having taken at least one dose of dabigatran prior to the event.

Exclusion criteria:

* Confirmed diagnosis of valvular AF (VAF);
* Documentation that the patient was taking dabigatran with other oral anticoagulant;
* Documentation of the patient receiving thrombolytic therapy prior to the event;
* Documentation that the patient was enrolled in an investigational clinical trial at the time of the event;
* Medical record was not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients with bleeding event using Dabigatran etexilate
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (22):
- United States (16):
  - Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - Boehringer Ingelheim Investigational Site, New Britain, Connecticut
  - Boehringer Ingelheim Investigational Site, Orlando, Florida
  - Boehringer Ingelheim Investigational Site, Tampa, Florida
  - Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, Hackensack, New Jersey
  - Boehringer Ingelheim Investigational Site, New York, New York
  - Boehringer Ingelheim Investigational Site, Staten Island, New York
  - Boehringer Ingelheim Investigational Site, Philedelphia, Pennsylvania
  - Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - Boehringer Ingelheim Investigational Site, Roanoke, Virginia
- Canada (6):
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational chart abstraction study.
Pre-assignment Details: 297 subjects were captured in the initial screening. 74 patients were deemed ineligible. A total of 3 patients were withdrawn after being included in the final study cohort following verification of ineligibility leaving 220 subjects eligible for study entry who were enrolled and included in the final study.
Groups:
- Dabigatran (Pradax® in Canada; Pradaxa® in the United States): Patients with Non-Valvular Atrial Fibrillation (NVAF) at two countries (United States and Canada) who received dabigatran etexilate (dabigatran capsules were approved at the 75 mg, 110 mg and 150 mg dosages, and the recommended dosing is orally twice daily).
Period: Overall Study
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States)
Started | 220
Completed | 220
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who received treatment at two countries (United States and Canada).
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States)
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.1 (10.3)
Gender [Count of Participants; unit: Participants]
  Female | 108
  Male | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Index Event Safety Outcomes (Ongoing/Resolved/Deceased) at Time of Hospital Discharge
Description: Percentages of patients with index event safety outcomes (ongoing/resolved/deceased) at the time of their hospital discharge/release.
  Emergency Department/Room (ED/ER).
  Bleeding status at the time of discharge were classified by the principal investigator, using medical record information and medical opinion, as:
  * Ongoing, if symptoms of bleeding not completely resolved at time of discharge;
  * Deceased in case of death;
  * Resolved otherwise.
Time Frame: From the time of presentation/admission to an ED/ER or hospitalization through all in-hospital referrals until discharge (between 28October2010 (the date of the first data entry)) and 01August2013 (the date of data entry closure); Up to 1008 days.
Population: Patients who received treatment at two countries (United States and Canada).
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States)
Number analyzed (Participants) | 220
Percentage of participants
  Ongoing | 19.1
  Resolved | 76.8
  Deceased | 4.1

2. Primary Outcome: Percentage of Patients Receiving Different Types of Interventions to Stop Index Events Until Hospital Discharge
Description: Percentages of patients receiving general intervention and general intervention combinations (i.e., medications, surgery, therapeutic procedures, transfusion/infusion, discontinuation of dabigatran) to manage the index events until their hospital discharge/release. Multiple interventions are possible.
Time Frame: From the time of presentation/admission to an ED/ER or hospitalization through all in-hospital referrals until discharge (between 28OCT2010 (the date of the first data entry)) and 01AUG2013 (the date of data entry closure); Up to 1008 days.
Population: Patients who received treatment at two countries (United States and Canada).
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States)
Number analyzed (Participants) | 220
Percentage of participants
  Any general intervention | 77.3
  Medications | 13.6
  Surgery | 6.8
  Therapeutic procedures | 9.5
  Transfusion/infusion | 36.8
  Discontinuation of dabigatran | 71.4
  No interventions | 22.7

3. Primary Outcome: Percentage of Bleeding Types and Anatomic Locations of the Index Event at Time of ED/ER Presentation
Description: Percentages of patients with index events by type (i.e. GI and/or GU) and anatomic location are presented. Multiple bleed locations are possible.
Time Frame: as for outcome 2
Population: Patients who received treatment at two countries (United States and Canada).
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States)
Number analyzed (Participants) | 220
Percentage of participants
  GI Bleed | 73.2
  Upper GI Bleed | 15.5
  Lower GI Bleed | 45.9
  GI Bleed - Location Unknown | 12.7
  GU Bleed | 28.6
  Both GI and GU | 0.2

ADVERSE EVENTS:
Time Frame: From the time of presentation/admission to an ED/ER or hospitalization through all in-hospital referrals until discharge: between 28October2010 (the date of the first data entry) and 01August2013 (the date of data entry closure); Up to 1008 days.
Description: As per the study protocol, the index gastrointestinal and/or and urogenital bleeding event leading to the inclusion of the patient in the study is also included in the definition of Adverse events (AEs).
Groups:
- Dabigatran (Pradax® in Canada; Pradaxa® in the United States: Patients with Non-Valvular Atrial Fibrillation (NVAF) at two countries (United States and Canada) who received dabigatran etexilate (dabigatran capsules were approved at the 75 mg, 110 mg and 150 mg dosages, and the recommended dosing is orally twice daily).
Arm/Group | Dabigatran (Pradax® in Canada; Pradaxa® in the United States
Serious Adverse Events (participants affected / at risk) | 184/220
Other Adverse Events (participants affected / at risk) | 79/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (Pradax® in Canada; Pradaxa® in the United States (N=220)
Haematuria (Renal and urinary disorders) | 32
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 52
Rectal haemorrhage (Gastrointestinal disorders) | 32
Anaemia (Blood and lymphatic system disorders) | 23
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 22
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 22
Haematochezia (Gastrointestinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Melaena (Gastrointestinal disorders) | 11
Atrial fibrillation (Cardiac disorders) | 4
Chest pain (General disorders) | 3
Dizziness (Nervous system disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 8
Hypotension (Vascular disorders) | 7
Nausea (Gastrointestinal disorders) | 2
Urinary tract infection (Infections and infestations) | 4
Cardiac failure congestive (Cardiac disorders) | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Anal haemorrhage (Gastrointestinal disorders) | 5
Haematemesis (Gastrointestinal disorders) | 6
Sepsis (Infections and infestations) | 6
Fatigue (General disorders) | 2
International normalised ratio increased (Investigations) | 3
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 3
Haemoglobin decreased (Investigations) | 4
Headache (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Syncope (Nervous system disorders) | 3
Tachycardia (Cardiac disorders) | 3
Urogenital haemorrhage (Renal and urinary disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Clostridium difficile infection (Infections and infestations) | 2
Coagulopathy (Blood and lymphatic system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Endocarditis (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Faeces discoloured (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Occult blood positive (Investigations) | 2
Orthostatic hypotension (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal failure (Renal and urinary disorders) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Ataxia (Nervous system disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Bladder obstruction (Renal and urinary disorders) | 1
Blood creatine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Calculus bladder (Renal and urinary disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Emphysematous cholecystitis (Infections and infestations) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
General physical condition abnormal (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Hemiparesis (Nervous system disorders) | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
International normalised ratio (Investigations) | 1
International normalised ratio abnormal (Investigations) | 1
International normalised ratio normal (Investigations) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Localised infection (Infections and infestations) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Microscopic polyangiitis (Vascular disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Renal atrophy (Renal and urinary disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urosepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (Pradax® in Canada; Pradaxa® in the United States (N=220)
Haematuria (Renal and urinary disorders) | 42
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 19
Rectal haemorrhage (Gastrointestinal disorders) | 26

LIMITATIONS AND CAVEATS:
Limitations of the data sources included completeness of information available in terms of potential lack of outcome data, medical history data and co-medications. Key limitations: 1. Generalizability. 2. Data quality. 3. Data availability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.